CLINICAL TRIAL: NCT02524743
Title: The Prevention of Pain Associated With Rocuronium Injection: Effect of Pretreatment With Acetaminophen and Lidocaine
Brief Title: The Prevention of Pain Associated With Rocuronium Injection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Filiz Alkaya Solmaz, Assistant Professor, MD, Suleyman Demirel University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 02.04.2014/48
Record Dates: First submitted 2015-08-05; First posted 2015-08-17 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-08

CONDITIONS: Injection Site Irritation
Keywords: Rocuronium; lidocaine; acetaminophen,; pain; injection
MeSH Terms: conditions — Pain | interventions — Acetaminophen; Lidocaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo (Group I) (Placebo Comparator): For pretreatment the patients were administered IV 5ml normal saline.
  A 20-gauge catheter was inserted into a superficial vein on the dorsum of the patient's non- dominant hand. The lactated Ringer's solution was infused at 100 ml/h for five minutes, The infusion was stopped and the arm with the IV line was elevated for 15 seconds for gravity drainage of venous blood. The venous drainage was occluded for 120 seconds by using a rubber tourniquet on the upper arm. During and after the injection of rocuromum, pain was graded with four point scale (TEST 1) and withdrawal movement was evaluated (TEST 2) by the study-blinded investigator
  Interventions: Other: Placebo
- Group II (Active Comparator): For pretreatment the patients were administered IV acetaminophen 50 mg
  A 20-gauge catheter was inserted into a superficial vein on the dorsum of the patient's non- dominant hand. The lactated Ringer's solution was infused at 100 ml/h for five minutes, The infusion was stopped and the arm with the IV line was elevated for 15 seconds for gravity drainage of venous blood. The venous drainage was occluded for 120 seconds by using a rubber tourniquet on the upper arm. During and after the injection of rocuromum, pain was graded with four point scale (TEST 1) and withdrawal movement was evaluated (TEST 2) by the study-blinded investigator
  Interventions: Drug: acetaminophen
- Group III (Active Comparator): For pretreatment the patients were administered IV acetaminophen 25 mg.
  A 20-gauge catheter was inserted into a superficial vein on the dorsum of the patient's non- dominant hand. The lactated Ringer's solution was infused at 100 ml/h for five minutes, The infusion was stopped and the arm with the IV line was elevated for 15 seconds for gravity drainage of venous blood. The venous drainage was occluded for 120 seconds by using a rubber tourniquet on the upper arm. During and after the injection of rocuromum, pain was graded with four point scale (TEST 1) and withdrawal movement was evaluated (TEST 2) by the study-blinded investigator
  Interventions: Drug: acetaminophen
- Group IV (Active Comparator): For pretreatment the patients were administered IV lidocaine 20 mg
  The venous drainage was occluded for 120 seconds by using a rubber tourniquet on the upper arm. During and after the injection of rocuromum, pain was graded with four point scale (TEST 1) and withdrawal movement was evaluated (TEST 2) by the study-blinded investigator
  Interventions: Drug: Lidocaine
- Group V (Active Comparator): For pretreatment the patients were administered IV lidocaine 40 mg.
  A 20-gauge catheter was inserted into a superficial vein on the dorsum of the patient's non- dominant hand. The lactated Ringer's solution was infused at 100 ml/h for five minutes, The infusion was stopped and the arm with the IV line was elevated for 15 seconds for gravity drainage of venous blood. The venous drainage was occluded for 120 seconds by using a rubber tourniquet on the upper arm. During and after the injection of rocuromum, pain was graded with four point scale (TEST 1) and withdrawal movement was evaluated (TEST 2) by the study-blinded investigator
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: acetaminophen — The venous drainage was occluded for 120 seconds by using a rubber tourniquet on the upper arm and the patients were pretreated acetaminophen (50mg and 25 mg IV) before the injection of rocuronium.Twenty seconds after the administration of rocuronium, 5 mg/kg of thiopental was administered IV. After orotracheal intubation, anesthesia was continued with sevofluorane during 40 % oxygen and 60 % air. Twenty-four hours after the operation, the injection site was checked for any complications, such as pain (absent/ present), swelling or allergic reaction by an anesthesiologist who did not know which drug was administered.
  Other Names: Parol; Perfalgan
  Arms: Group II; Group III
Drug: Lidocaine — The venous drainage was occluded for 120 seconds by using a rubber tourniquet on the upper arm and the patients were pretreated lidocaine (20 mg and 40 mg IV) before the injection of rocuronium.Twenty seconds after the administration of rocuronium, 5 mg/kg of thiopental was administered IV. After orotracheal intubation, anesthesia was continued with sevofluorane during 40 % oxygen and 60 % air. Twenty-four hours after the operation, the injection site was checked for any complications, such as pain (absent/ present), swelling or allergic reaction by an anesthesiologist who did not know which drug was administered.
  Other Names: Aritmal % 2; Jetmonal %10
  Arms: Group IV; Group V
Other: Placebo — The venous drainage was occluded for 120 seconds by using a rubber tourniquet on the upper arm and the patients were pretreated 5 ml iv normal saline before the injection of rocuronium.Twenty seconds after the administration of rocuronium, 5 mg/kg of thiopental was administered IV. After orotracheal intubation, anesthesia was continued with sevofluorane during 40 % oxygen and 60 % air. Twenty-four hours after the operation, the injection site was checked for any complications, such as pain (absent/ present), swelling or allergic reaction by an anesthesiologist who did not know which drug was administered.
  Other Names: Saline
  Arms: Placebo (Group I)

SUMMARY:
The purpose of this study is to determine whether efficacy of different doses of lidocain and acetaminophen for the prevention of rocuronium injection pain and frequency of withdrawal movements during the general anesthesia induction period.

DETAILED DESCRIPTION:
The study was conducted on 150 patients aged 18- 70 years of ASA (American Society of Anesthesiologists) physical status I- II who were to undergo various elective operations. None of the patients was premedicated before the operation. The patients were monitored with three derivation electrocardiogram, non- invasive arterial pressure, and pulse oximeter.

A 20-gauge catheter was inserted into a superficial vein on the dorsum of the patient's non- dominant hand. The lactated Ringer's solution was infused at 100 ml/h for five minutes, The infusion was stopped and the arm with the IV line was elevated for 15 seconds for gravity drainage of venous blood, The venous drainage was occluded for 120 seconds by using a rubber tourniquet on the upper arm and the patients were pretreated by either lidocaine (20 mg and 40 mg IV) or acetaminophen (50mg and 25 mg IV) before the injection of rocuronium. Some patients received 5 ml normal saline. The patients were randomly assigned to five groups. For pretreatment the patients were administered 5 ml normal saline in Group I (Control); acetaminophen 50mg in Group II, acetaminophen 25 mg in Group III, lidocaine 20 mg in Group IV and lidocaine 40mg in Group V, diluted into 5 mL of saline IV. The occlusion was released after 120 s and 0.6 mg/kg of rocuronium 1% was injected IV over 5 seconds. During and after the injection of rocuronium, pain was graded with four point scale (TEST 1) and withdrawal movement was evaluated (TEST 2) by the study-blinded investigator. Twenty seconds after the administration of rocuronium, 5 mg/kg of thiopental was administered IV. After orotracheal intubation, anesthesia was continued with sevofluorane during 40 % oxygen and 60 % air. Twenty-four hours after the operation, the injection site was checked for any complications, such as pain (absent/ present), swelling or allergic reaction by an anesthesiologist who did not know which drug was administered.

Table 1: Four Point Scala (TEST 1) Degree of pain Response Pain score

1. None: Negative response to questioning: 0
2. Mild: Pain reported in response to questioning only, without any behavioral signs: 1
3. Moderate: Pain reported in response to questioning and accompanied by a behavioral sign, or pain reported spontaneously without questioning: 2
4. Severe: Strong vocal response or response accompanied by facial grimacing, arm withdrawal, or tears : 3

Table 2: Evaluation Of Withdrawal Movements During Rocuronium Injection ( TEST2) Pain Score Response

1. No response
2. Movement at wrist only
3. Movement/ withdrawal involving arm only (elbow/ shoulder)
4. Generalized response ( movement/ withdrawal in more than one extremity, cough or breath holding)

ELIGIBILITY:
Inclusion Criteria:

* 18- 70 years of ASA physical status I- II who were to undergo various elective operations.

Exclusion Criteria:

* Patients with chronic pain syndrome,
* Patients with neurologic deficits,
* Patients with thrombophlebitis,
* Patients with difficult venous access,
* Patients with allergy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2014-05; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Change in intraoperative pain | 10 seconds
  pain was graded with four point scale (TEST 1) and withdrawal movement was evaluated (TEST 2)

SECONDARY OUTCOMES:
Change in postoperative pain | 24 hours
  Twenty-four hours after the operation, the injection site was checked for any complications, such as pain, swelling or allergic reaction

CONTACTS AND LOCATIONS:
Overall Officials: Filiz Alkaya Solmaz, Principal Investigator — Suleyman Demirel University Hospital

REFERENCES:
- [Background] Steegers MA, Robertson EN. Pain on injection of rocuronium bromide. Anesth Analg. 1996 Jul;83(1):203. doi: 10.1097/00000539-199607000-00065. No abstract available. PMID 8659757
- [Background] Kwak HJ, Kim JY, Kim YB, Min SK, Moon BK, Kim JY. Pharmacological prevention of rocuronium-induced injection pain or withdrawal movements: a meta-analysis. J Anesth. 2013 Oct;27(5):742-9. doi: 10.1007/s00540-013-1595-7. Epub 2013 Mar 22. PMID 23519582
- See also: Springer — http://link.springer.com/article/10.1007%2Fs00540-013-1595-7